CLINICAL TRIAL: NCT05769062
Title: Identification and Prevention of Pelvic Floor Dysfunction in Gynecologic Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Former PI left the institution so enrollment was closed early.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202209105
Record Dates: First submitted 2023-02-16; First posted 2023-03-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Gynecologic Cancer
Keywords: cervical cancer; radiation; chemoradiation; pelvic floor muscle dysfunction; chronic pelvic pain
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-digit pelvic exam (Experimental): * Patients will have a pelvic floor muscle exam performed by their gynecologic radiation oncologist prior to treatment, at treatment mid-point (after 3 weeks of treatment), at the end of treatment (after 6 weeks of treatment), and at a follow-up visit 6 months after the end of treatment. Patients will also complete the Pelvic Floor Impact Questionnaire 7 (PFIQ-7), Pelvic Floor Disability Index (PFDI-20), and the EORTC QLQ-CX24 at these time points.
  * The patient will also undergo a standard of care MRI prior to starting treatment.
  Interventions: Procedure: Single digit pelvic exam

INTERVENTIONS:
Procedure: Single digit pelvic exam — The exam takes approximately 5 minutes and uses a single digit to palpate the pelvic floor muscles, during which patients will rate pain on a scale of 0-10 at 5 paired locations.

SUMMARY:
The two goals of this study are to establish a standardized method of assessing the pelvic floor for patients undergoing pelvic radiation and to determine the feasibility of inverse-RT planning using MRI to identify dosimetric constraints of the pelvic floor musculature for use in radiation planning. The investigators hypothesize that an exam-based diagnostic tool will provide more information about the areas of injury related to pelvic radiation than patient-reported outcomes, and could be used in future studies of preventive strategies. An exam-based tool will also allow measurement of the pain dose-response to radiation treatment of specific areas, which could be excluded from radiation fields during treatment planning.

ELIGIBILITY:
Inclusion Criteria - Prospective Cohort

* Undergoing primary treatment for locally advanced cervical cancer with definitive, curative-intent chemoradiotherapy (chemotherapy must be a radiosensitizing platinum agent).
* At least 18 years of age.
* English speaker.
* Able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria - Prospective Cohort

* Received any form of pelvic radiation (excepting diagnostic studies).
* Currently taking and does not plan to take anti-estrogenic hormonal therapy.
* Diagnosis of interstitial cystitis/chronic bladder pain, irritable bowel syndrome, or inflammatory bowel disease.
* Currently being treated for a chronic non-cancer pain condition (treatment for pain after enrollment is acceptable).

Inclusion Criteria - Retrospective Cohort (historical control)

* Received primary treatment for locally advanced cervical cancer with definitive, curative-intent chemoradiotherapy (chemotherapy must be a radiosensitizing platinum agent).
* At least 18 years of age.

Exclusion Criteria - Retrospective Cohort (historical control)

* Received any form of pelvic radiation (excepting diagnostic studies).
* Took anti-estrogenic hormonal therapy during treatment or in the 6 months following treatment.
* Diagnosis of interstitial cystitis/chronic bladder pain, irritable bowel syndrome, or inflammatory bowel disease at the start of treatment.
* Simultaneously treated for a chronic non-cancer pain condition at the start of treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Comparison of patient-reported symptoms as measured by EORTC QLQ-CX2 compared to findings of single digit pelvic exam | Prior to starting treatment, at treatment mid-point (3 weeks after treatment), at end of treatment (after 6 weeks of treatment), and at 6 month follow-up visit after end of treatment
  An exam will be considered positive for PFMD if pain at any examined site is reported as greater than or equal to four (>4) out of 10. The EORTC QLQ-CX2 contains 24 items scored 1-4 by frequency with which the patient experiences each. The minimum possible score is 24, and maximum 96, with higher scores indicating worse quality of life. The questionnaire will be considered positive if any vaginal, sexual, or genitourinary module question is rated 4 and otherwise will be analyzed as a continuous variable.
Comparison of patient-reported symptoms as measured by PFDI-20 compared to findings of single digit pelvic exam | Prior to starting treatment, at treatment mid-point (3 weeks after treatment), at end of treatment (after 6 weeks of treatment), and at 6 month follow-up visit after end of treatment
  An exam will be considered positive for PFMD if pain at any examined site is reported as >4 out of 10. The PFDI-20 includes 20 items in three domains and provides a scaled score of 0-100 indicating how much a patient is bothered by pelvic floor-related issues. The questionnaire will be considered positive if the scaled score is greater than or equal to 16, indicating at least "moderate distress" and otherwise will be analyzed as a continuous variable.
Comparison of patient-reported symptoms as measured by PFIQ-7 compared to findings of single digit pelvic exam | Prior to starting treatment, at treatment mid-point (3 weeks after treatment), at end of treatment (after 6 weeks of treatment), and at 6 month follow-up visit after end of treatment
  An exam will be considered positive for PFMD if pain at any examined site is reported as >4 out of 10. The PFIQ-7 includes 7 items each repeated across three domains and provides a scaled score and total score indicating how much a patient is bothered by pelvic floor-related issues. The questionnaire does not have an established severity scale, and therefore will be analyzed as a simple continuous variable.

SECONDARY OUTCOMES:
Time course of pelvic floor dysfunction evolution over the course of treatment for cervical cancer using pelvic exam | Through completion of follow-up (estimated to be 6 months)
  Continuous variables of scales and total scores will be calculated for the exam at each time point and represented in spider-type plots. Results of the exam will be analyzed using the thresholds described in the primary outcome measure, and frequencies of positive scores reported for each time point.
Time course of pelvic floor dysfunction evolution over the course of treatment for cervical cancer using the EORTC QLQ-CX2 scores | Through completion of follow-up (estimated to be 6 months)
  Continuous variables of scales and total scores will be calculated for the questionnaires at each time point and represented in spider-type plots. Results of the questionnaire will be analyzed using the thresholds described in the primary outcome measure, and frequencies of positive scores reported for each time point.
Time course of pelvic floor dysfunction evolution over the course of treatment for cervical cancer using the PFDI-20 scores | Through completion of follow-up (estimated to be 6 months)
  Continuous variables of scales and total scores will be calculated for the questionnaires at each time point and represented in spider-type plots. Results of the questionnaire will be analyzed using the thresholds described in the primary outcome measure, and frequencies of positive scores reported for each time point.
Time course of pelvic floor dysfunction evolution over the course of treatment for cervical cancer using the PFIQ-7 scores | Through completion of follow-up (estimated to be 6 months)
  Continuous variables of scales and total scores will be calculated for the questionnaires at each time point and represented in spider-type plots. Results of the questionnaire will be analyzed using the thresholds described in the primary outcome measure, and frequencies of positive scores reported for each time point.
Correlate radiation dose to pelvic floor structures with symptom severity by questionnaire (EORTC QLQ-CX2, PFDI-20, and PFIQ-7) and physical exam | Through completion of follow-up (estimated to be 6 months)
  Continuous variables of scales and total scores, as well as specific scores for radiation-exposed structures on exam, will be compared to dosimetric assessments of exposure of pelvic floor structures.
Determine structure level radiation dose to complex functional pelvic structures | Through completion of follow-up (estimated to be 6 months)
  Standard dosimetric values will be calculated for each specific pelvic floor structure evaluated on exam.
Frequency of pelvic floor muscle dysfunction symptoms in split-field IMRT patients compared to historical controls | Through completion of follow-up (estimated to be 6 months)
  Historical controls will be queried via chart review for dosimetric values in archived radiation treatment plans and compared to current gynecologic radiation standards. These patients will also undergo thorough chart review for subsequent diagnoses of pelvic floor-related disorders and compared to the diagnosis rate using the proposed screening tools in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Premal Thaker, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu